CLINICAL TRIAL: NCT02566057
Title: Prospective Pharmacogenetic Testing and Clinical Outcomes in Patients With Early-Phase Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Genomind, LLC (Industry)
Responsible Party: Principal Investigator, Jianping Zhang, Psychiatrist, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-587B
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder; Psychotic Disorders; Bipolar Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PGx testing guided treatment (PGT) (Experimental): Results of the GeneceptTM Assay will be provided to their prescribers who may use the knowledge to guide medication management.
  Interventions: Biological: PGx testing guided treatment (PGT)
- Treatment as usual condition (TAU) (No Intervention): Patients will also utilize the GeneceptTM Assay but the results will not be provided back to their prescribers, who will treat the patients without the knowledge of pharmacogenetic testing results.

INTERVENTIONS:
Biological: PGx testing guided treatment (PGT) — Genecept Assay (GeneceptTM Assay) will provide information on genotypes of genetic variants that are relevant to psychiatric drug response. The provider can use the information to decide on which psychotropic drugs to use.
  Arms: PGx testing guided treatment (PGT)

SUMMARY:
This study evaluates whether prospective pharmacogenetic testing is cost-effective in affecting clinical treatment outcomes in patients with early-phase psychosis.

DETAILED DESCRIPTION:
Large scale clinical trials have demonstrated that a substantial proportion of patients with psychotic disorders, such as schizophrenia and bipolar disorder, discontinue their antipsychotic medications due to either lack of efficacy or intolerable side effects, such as extrapyramidal symptoms (EPS) and weight gain. In clinical practice, it is essentially a trial and error process in deciding the best antipsychotic drug to start or switch to after a failed trial as there is little empirical data available to guide clinicians in drug selection. One promising tool, which can potentially provide valuable information to help guide medication management, is pharmacogenetic testing of certain genetic variants that are associated with psychiatric drug response. However, most pharmacogenetic studies to date have been retrospective, and there is no prospective clinical trial evaluating the clinical utility of pharmacogenetic testing in guiding clinical practice. Furthermore, it is unknown whether pharmacogenetic testing is cost effective.

Until recently, pharmacogenetic testing has been expensive and time-consuming. New technology in the past few years makes it possible for cheaper and faster testing. One of the companies that offer pharmacogenetic testing services, Genomind LLC, provides genotyping of variants (GeneceptTM Assay) that are relevant to psychiatric drug response. For example, the serotonin 2C receptor gene (HTR2C) has variants that protect patients from antipsychotic drug induced weight gain (-759C/T, rs3813929); a deletion variant of the dopamine D2 receptor gene (DRD2) suggests poor efficacy with antipsychotic drug treatment (-141C Ins/Del, rs1799732); the short allele of the serotonin transporter gene (SLC6A4) is associated with antidepressant side effects.

In the present study, investigators propose to conduct a prospective, randomized, rater-blinded clinical trial to test the clinical utility and cost-effectiveness of pharmacogenetic testing in guiding medication treatment in patients with recent-onset psychotic disorders. Patients will be assigned to either a pharmacogenetic testing guided treatment condition (PGT) or a treatment as usual condition (TAU). In the PGT condition, patients will utilize the GeneceptTM Assay and results will be provided to their prescribers who may use the results to guide medication management. In the TAU condition, patients will also utilize the GeneceptTM Assay but the results will not be provided back to their prescribers, who will treat the patients without the knowledge of pharmacogenetic testing results.

Pharmacogenetic testing may be more relevant in recent-onset or early stage illnesses because past medication history that is typically used to guide medication choice may not be available. Pharmacogenomic testing may be particularly pertinent to younger patients because they tend to be medication naïve and do not have previous medication history to guide future treatment. Pharmacogenomic testing may provide valuable information to guide medication choice in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age 15-64;
2. Diagnostic and Statistical Manual Diploma in Social Medicine diagnosis of schizophrenia (DSM IV), schizoaffective disorder, schizophreniform disorder, psychotic disorder NOS, and bipolar disorder;
3. Onset of antipsychotic treatment within the past 3 years;
4. Able to provide informed consent. (assent for those under age 18)

Exclusion Criteria:

1. Evidence of serious medical conditions,
2. Female patients who are pregnant or breast feeding;
3. Patients who are not willing to take medications for treatment;
4. Patients who are unable to provide informed consent due to impairment in decision-making ability.

Ages: 15 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2014-07-10 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Time to Discontinuation of First Medication | 12 months
  Due to lack of efficacy or intolerability

SECONDARY OUTCOMES:
Prescribing Behavior Change Based on the Results of the Pharmacogenetic Testing | 12 months
  The clinician is asked to fill out a questionnaire elaborating the medication decision-making process for each patient, including whether or not acting on the genetic information provided clinically relevant information.

OTHER OUTCOMES:
Treatment Efficacy | 12 months
  Assessed by Brief Psychiatric Rating Scale (BPRS)
Adverse Drug Response | 12 months
  Assessed by measures including Hillside Adverse Events Rating Scale (HAERS), Simpson-Angus Rating Scale for Extrapyramidal Symptoms (SARSES), Barnes Rating Scale for Drug-Induced Akathisia (BRSDIA), Abnormal Involuntary Movement Scale (AIMS)
Treatment Services Utilized | 12 months
  Examine overall medical costs (including outpatient visits, procedures, hospitalizations, other professional charges, laboratory charges, and medication costs), as well as costs specifically associated with treatment of psychiatric symptoms based upon ICD9 code (for procedures and visits) and medication category. This information will be provided by insurance company for patients with ValueOptions insurance coverage.

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Zhang, MD, PhD, Principal Investigator — Psychiatrist
Locations (1):
- Zucker Hillside Hospital-North Shore Long Island Jewish Health System, Glen Oaks, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malhotra AK, Zhang JP, Lencz T. Pharmacogenetics in psychiatry: translating research into clinical practice. Mol Psychiatry. 2012 Jul;17(8):760-9. doi: 10.1038/mp.2011.146. Epub 2011 Nov 15. PMID 22083729
- [Background] Zhang JP, Malhotra AK. Pharmacogenetics and antipsychotics: therapeutic efficacy and side effects prediction. Expert Opin Drug Metab Toxicol. 2011 Jan;7(1):9-37. doi: 10.1517/17425255.2011.532787. PMID 21162693